CLINICAL TRIAL: NCT04617548
Title: Feasibility Testing of tDCS and Metacognitive Strategy Training in Chronic Stroke
Brief Title: tDCS and CO-OP in Chronic Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Anna Boone, Anna E. Boone, MSOT, PhD, OTR/L, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009451
Record Dates: First submitted 2020-09-25; First posted 2020-11-05 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Chronic Stroke
Keywords: Stroke; Metacognitive Strategy Training; Brain Stimulation; CO-OP; tDCS
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- tDCS and CO-OP Group (Experimental): One-hour session three times per week for 4 weeks. Participants will receive anodal tDCS (1.5 mA) to the dorsolateral prefrontal cortex (dlPFC) for 20 minutes at the beginning of each session. Following each tDCS session, the participants will complete a sensations questionnaire.The basis for each session will be task-based practice of client-chosen goals and the use of cognitive strategies using CO-OP.
  Interventions: Combination Product: tDCS and CO-OP Group

INTERVENTIONS:
Combination Product: tDCS and CO-OP Group — Transcranial direct current stimulation modulates the excitability of targeted brain regions, and is thought to facilitate or inhibit neuroplasticity. Participants will receive anodal tDCS (1.5 mA) to the dorsolateral prefrontal cortex (dlPFC) for 20 minutes at the beginning of each session. CO-OP focuses on learning of a global problem-solving strategy, Goal-Plan-Do-Check (GPDC), within the performance of participant-chosen goals. Use of a broadly applicable strategy and meaningful activity ensures the intervention is salient to the participant and increases likelihood of transfer. Uniquely, therapists applying CO-OP use guided discovery methods to support participants in analyzing their own performance of a given task and generating potential solutions for improving performance. Participants become equipped with these skills through repetitive application of the Goal-Plan-Do-Check process.The intervention focuses on learning GPDC with gradual withdrawal of guided discovery methods.
  Other Names: Brain Stimulation and Metacognitive Strategy

SUMMARY:
This project seeks to evaluate the acceptability feasibility, practicality feasibility, and preliminary effect of combining transcranial direct current stimulation (tDCS) and metacognitive strategy training (MCST) in individuals with chronic stroke.

DETAILED DESCRIPTION:
Currently seven million people are living in the United States post stroke, making stroke the leading cause of long term disability. Almost half of the people living in the community following stroke have problems that challenge the activities that support their daily lives. This is in part due to the rehabilitation community's focus on short term stroke recovery and not on supporting survivors' need to actively manage their long-term disability and the environment around them so they can return to full participation in communities of their choice post-rehabilitation. The rehabilitation community is in need of evidence-based interventions for addressing post-stroke functional limitations. Metacognitive strategy training is a performance-based, problem-solving approach to task performance difficulties. Participants are taught to identify when to apply a cognitive strategy, how to apply it, and how to monitor and adapt usage of cognitive strategies within task performance. Metacognitive strategy training is recognized as a practice standard for addressing functional limitations post-stroke. Transcranial direct current stimulation is a method that has been used for over 15 years to modulate the excitability of targeted brain regions. While it does not directly stimulate neurons, it results in changes to polarity of neuronal membranes and is thought to facilitate or inhibit neuroplasticity. Combination of these approaches may result in an interaction of effects and a greater effect on function in individuals post-stroke than either approach used alone.

ELIGIBILITY:
Inclusion Criteria:

* > 6 months post mild to moderate ischemic stroke
* self-reported functional limitations
* Age 30-80

Exclusion Criteria:

* history of other neurological diagnoses
* cognitive impairment (less than or equal to 21 on the Montreal Cognitive Assessment)
* severe aphasia (greater than or equal to 2 on the NIHSS language item
* non-English speaking
* any additional condition where the PI deems participation unsafe
* pregnancy, 7)
* history of seizures
* medications that influence cortical excitability
* metallic implants above the chest
* history of welding or metalwork
* severe depressive symptoms (>21 on Patient Health Questionnaire)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), & Feasibility of Intervention Measure | after study completion, an average of 5 weeks
  A brief questionnaire to evaluate participant satisfaction regarding the intervention's acceptability, appropriateness, and feasibility
Semi-Structured Interview | after study completion, an average of 5 weeks
  A brief interview to gather participant perceptions of the intervention, including their perceived benefit and practicality of the intervention and suggestions for improvement for the intervention.
Client Satisfaction Questionnaire (CSQ-8) | after study completion, an average of 5 weeks
  Self-report, 8 item measures of intervention acceptability

SECONDARY OUTCOMES:
Performance Quality Rating Scale (PQRS) | Pre-intervention and post-intervention, typically an average of 5 weeks
  An objective measure of participant performance of goals. Each goal is rated by a trained observer from 1 (no activity criteria were met) and 10 (all activity criteria were met).
Canadian Occupational Performance Measure (COPM) | Pre-intervention and post-intervention, typically an average of 5 weeks
  Self-report measures of perceived performance and satisfaction of occupational performance on a 1 to 10 Likert scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cicerone KD, Langenbahn DM, Braden C, Malec JF, Kalmar K, Fraas M, Felicetti T, Laatsch L, Harley JP, Bergquist T, Azulay J, Cantor J, Ashman T. Evidence-based cognitive rehabilitation: updated review of the literature from 2003 through 2008. Arch Phys Med Rehabil. 2011 Apr;92(4):519-30. doi: 10.1016/j.apmr.2010.11.015. PMID 21440699
- [Background] Hartman-Maeir A, Soroker N, Ring H, Avni N, Katz N. Activities, participation and satisfaction one-year post stroke. Disabil Rehabil. 2007 Apr 15;29(7):559-66. doi: 10.1080/09638280600924996. PMID 17453976
- [Background] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425
- [Background] Liebetanz D, Koch R, Mayenfels S, Konig F, Paulus W, Nitsche MA. Safety limits of cathodal transcranial direct current stimulation in rats. Clin Neurophysiol. 2009 Jun;120(6):1161-7. doi: 10.1016/j.clinph.2009.01.022. Epub 2009 Apr 28. PMID 19403329
- [Background] McEwen S, Polatajko H, Baum C, Rios J, Cirone D, Doherty M, Wolf T. Combined Cognitive-Strategy and Task-Specific Training Improve Transfer to Untrained Activities in Subacute Stroke: An Exploratory Randomized Controlled Trial. Neurorehabil Neural Repair. 2015 Jul;29(6):526-36. doi: 10.1177/1545968314558602. Epub 2014 Nov 21. PMID 25416738
- [Background] Nitsche MA, Liebetanz D, Lang N, Antal A, Tergau F, Paulus W. Safety criteria for transcranial direct current stimulation (tDCS) in humans. Clin Neurophysiol. 2003 Nov;114(11):2220-2; author reply 2222-3. doi: 10.1016/s1388-2457(03)00235-9. No abstract available. PMID 14580622
- [Background] Paulus W. Outlasting excitability shifts induced by direct current stimulation of the human brain. Suppl Clin Neurophysiol. 2004;57:708-14. doi: 10.1016/s1567-424x(09)70411-8. PMID 16106673
- [Background] Polania R, Nitsche MA, Paulus W. Modulating functional connectivity patterns and topological functional organization of the human brain with transcranial direct current stimulation. Hum Brain Mapp. 2011 Aug;32(8):1236-49. doi: 10.1002/hbm.21104. Epub 2010 Jul 6. PMID 20607750
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Richards LG, Latham NK, Jette DU, Rosenberg L, Smout RJ, DeJong G. Characterizing occupational therapy practice in stroke rehabilitation. Arch Phys Med Rehabil. 2005 Dec;86(12 Suppl 2):S51-S60. doi: 10.1016/j.apmr.2005.08.127. PMID 16373140